CLINICAL TRIAL: NCT02530671
Title: Effect of a Multi-directional Power and a Manual Toothbrush in Subjects Susceptible to Gingival Recession: A 12-month Randomized Controlled Clinical Study
Brief Title: Effect of a Multi-directional Power Toothbrush on Recession
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Principal Investigator, Sonja Sälzer, Dr. Sonja Sälzer, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2011015
Record Dates: First submitted 2015-08-18; First posted 2015-08-21 (Estimated); Results first posted 2015-10-19 (Estimated); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Gingival Recession
Keywords: multi-directional power toothbrush; manual toothbrush
MeSH Terms: conditions — Gingival Recession | interventions — Toothbrushing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual toothbrush (Active Comparator): ADA reference manual toothbrush
  Interventions: Device: Toothbrushing with manual toothbrush
- Power toothbrush (Experimental): Multi-directional power toothbrush
  Interventions: Device: Toothbrushing with power toothbrush

INTERVENTIONS:
Device: Toothbrushing with manual toothbrush
  Arms: Manual toothbrush
Device: Toothbrushing with power toothbrush
  Arms: Power toothbrush

SUMMARY:
Background: Clinical studies have explored the relationship between toothbrushing and the development of recession, but relevant recession data for the multi-directional power toothbrush (PT) are lacking. The aim of this study was to evaluate the effect of brushing with either a multi-directional power toothbrush (PT) or an ADA (American Dental Association) reference manual toothbrush (MT) on pre-existing mid-buccal gingival recession (Pre-GR) over 12 months

Methods: This was a 12-month, prospective, single-blind, parallel-group, randomized controlled clinical study. Healthy participants without periodontitis but with at least 2 teeth showing Pre-GR ≥2mm were randomized to a group either brushing with a MT or a PT. The primary outcome parameter was the change at sites with Pre-GR ≥2mm. All recession measurements were performed by one calibrated examiner at baseline, 6 and 12 months. Secondary outcomes were changes of recession at all buccal sites (with or without pre-GR), changes in the percentage of recession sites demonstrating a change of ≥1mm as well as changes in pocket probing depths.

ELIGIBILITY:
Inclusion Criteria:

* 18 scorable teeth without orthodontic appliances or crowns and bridges
* at least 2 teeth showing recession of ≥ 2 mm on the mid-buccal surfaces (high risk teeth)

Exclusion Criteria:

* evidence of neglected dental health
* periodontitis and/or major hard/soft tissue lesions
* any physical limitations or restrictions potentially interfering with normal oral hygiene
* therapy with any drug within 28 days prior to the study
* pregnancy or breast feeding
* any systematic condition or significant illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2014-06 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Manual Toothbrush: ADA (American Dental Association) reference manual toothbrush
  Toothbrushing with manual toothbrush
- Power Toothbrush: Multi-directional power toothbrush
  Toothbrushing with power toothbrush
Period: Overall Study
Arm/Group | Manual Toothbrush | Power Toothbrush
Started | 55 | 55
Completed | 52 | 55
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Manual Toothbrush: ADA reference manual toothbrush
  Toothbrushing with manual toothbrush
- Total: Total of all reporting groups
Arm/Group | Manual Toothbrush | Power Toothbrush | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (9.7) | 32 (12.5) | 31 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 31 | 63
  Male | 23 | 24 | 47
Region of Enrollment [Number; unit: participants]
  Germany | 55 | 55 | 110
Smoker (Yes/Now) [Number; unit: participants]
  Yes | 7 | 7 | 14
  No | 48 | 48 | 96
Previous used toothbrush (MT/PT) [Number; unit: participants]
  Manual Toothbrush | 40 | 27 | 67
  Power Toothbrush | 15 | 28 | 43

OUTCOME MEASURES:

1. Primary Outcome: Gingival Recession at Sites With Preexisting Recessions ≥2mm
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Manual Toothbrush | Power Toothbrush
Number analyzed (Participants) | 55 | 55
mm | 2.09 (0.29) | 2.08 (0.30)

2. Secondary Outcome: Recession at All Buccal Sites
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Manual Toothbrush | Power Toothbrush
Number analyzed (Participants) | 55 | 55
mm | 0.416 (0.18) | 0.007 (0.16)

3. Secondary Outcome: Percentage of Recession Sites Demonstrating a Change of ≥1mm
Time Frame: 12 months
Measure: Number; unit: percentage of sites
Arm/Group | Manual Toothbrush | Power Toothbrush
Number analyzed (Participants) | 55 | 55
percentage of sites
  decrease | 14 | 24
  increase | 9 | 5

4. Secondary Outcome: Pocket Probing Depths at 12months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Manual Toothbrush | Power Toothbrush
Number analyzed (Participants) | 55 | 55
mm | 1.91 (0.17) | 1.88 (0.18)

5. Primary Outcome: Bristle Splay Index (BSI) After a Specific Time-of-use
Description: A digital computer program (ImageJ, NIH, Bethesda, MD, USA) for evaluating the index was applied. All brushes were photographed from both top and side view in a standardized set-up including a benchmark (Lego GmbH (Gemeinschaft mit beschränkter Haft), Grasbrunn, Germany) as reference for measurement. Subsequently, an independent examiner (N.H.) measured the lengths twice. To devise the BSI formula the results were averaged and inserted. The formula is defined by: BSI (%) = ((a´- a)/a + (b´- b)/b + (c´- c)/c + (d´- d)/d)/4 x 100. BSI was standardized for usage time by dividing it by the number of days used (BSI/T).
Time Frame: 3, 6, 9 and 12 months
Measure: Mean (Standard Deviation); unit: percentage of the original bristle field
Arm/Group | Manual Toothbrush | Power Toothbrush
Number analyzed (Participants) | 55 | 54
percentage of the original bristle field | 0.2 (0.2) | 0.1 (0.1)

6. Secondary Outcome: Comparison of BSI Between Periods
Time Frame: 0-3, 9-12 months
Measure: Mean (Standard Deviation); unit: percentage of the original bristle field
Arm/Group | Manual Toothbrush | Power Toothbrush
Number analyzed (Participants) | 54 | 55
percentage of the original bristle field
  0-3 months | 23.6 (14) | 6.4 (11)
  9-12months | 28.0 (14.8) | 9.8 (12.1)

ADVERSE EVENTS:
Arm/Group | Manual Toothbrush | Power Toothbrush
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No